CLINICAL TRIAL: NCT05662358
Title: Denosumab vs Alendronate in Patients With Osteoporotic Vertebral Compression Fracture After Percutaneous Vertebroplasty: A Randomized Controlled Trial
Brief Title: Denosumab vs Alendronate After Vertebroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShenzhenPH06
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Denosumab Allergy
MeSH Terms: interventions — Denosumab; Injections, Subcutaneous; Alendronate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): 1 ml (60 mg) of denosumab (Prolia; Amgen, Inc) subcutaneous injection plus intravenous placebo every 6 months
  Interventions: Drug: Denosumab; Drug: Placebo
- alendronate (Active Comparator): oral 70 mg alendronate sodium weekly.
  Interventions: Drug: Alendronate; Drug: Placebo

INTERVENTIONS:
Drug: Denosumab — 1 ml (60 mg) of denosumab (Prolia; Amgen, Inc) subcutaneous injection
  Other Names: Denosumab 6 month/subcutaneous
  Arms: Denosumab
Drug: Alendronate — oral 70 mg alendronate sodium weekly plus subcutaneous placebo per 6 month.
  Other Names: oral alendronate
  Arms: alendronate
Drug: Placebo — oral placebo weekly

SUMMARY:
Osteoporotic vertebral compression fracture (OVCF) patients had a proportion of secondary fractures after percutaneous vertebroplasty (PVP). Denosumab and alendronate is both effective to prevent bone loss for OVCF postmenopausal women. However, trial evidence comparing effect of denosumab vs zoledronate after PVP was unknown. The study aims to assess the efficiency of denosumab vs alendronate for OVCF patients bone mineral density (BMD), bone turnover markers (BTMs), secondary fracture and adverse events after PVP

DETAILED DESCRIPTION:
Whether denosumab was non-inferior than alendronate in improving bone mineral density (BMD), bone turnover markers (BTMs), functional status questionnaires, and secondary fracture in elderly patients with OVCF after PVP remains unknown. A prospective, randomized, placebo-controlled clinical trial in OVCF patients with PVP was performed. This study aimed to investigate the efficiency of denosumab vs alendronate on BMD, BTMs, functional status, secondary fracture rate, and adverse events in OVCF patients after PVP during a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Must be age between 50 and 85 years old

  * X-ray diagnosis of 1 or 2 segment vertebral compression fractures from T4 to L5
  * Bone mineral density T value less than -1 via dual-energy X-ray
  * A recent fracture history less than 6 weeks
  * MRI show bone marrow edema of fractured vertebrae
  * low back pain, local paravertebral tenderness

Exclusion Criteria:

* Must be able to have no intervertebral fissure

  * Must be able to have no infection
  * Must be able to have no malignancy
  * Must be able to have no neurological dysfunction
  * Must be able to have no previous use of anti-osteoporosis drugs
  * Must be able to have no inability to perform magnetic resonance imaging
  * Must be able to have no prior back open surgery
  * Must be able to have no other established contraindications for elective surgery

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Lumbar bone mineral density(BMD) | up to 12 months
  Lumbar vertebral (L1 to L4, except the surgery segment) BMD were determined at baseline, 6 and 12 months via dual energy X-ray
Total hip BMD | up to 12 months
  Total hip BMD were determined at baseline, 6 and 12 months via dual-energy X-ray.
Femoral neck BMD | up to 12 months
  Femoral neck BMD were determined at baseline, 6 and 12 month via dual-energy X-ray
Procollagen type 1 n-terminal propeptide (P1NP) | up to 12 months
  Bone formation marker, P1NP were determined at baseline, 6 and 12 months after surgery.
C-terminal cross-linked type 1 collagen terminal peptide (CTX) | up to 12 months
  Bone resorption marker, CTX were determined at baseline, 6 and 12 months after surgery
Visual analog scale (VAS) back | up to 12 months
  The VAS score for back pain were determined at baseline, 6 and 12 month. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is scored by 24 adding up the number of items checked "yes" on different low back pain-related daily activity disabilities. Total scores range from 0 to 24, with higher scores 24 indicating a higher level of disability related to low back pain and lowest 0 represents no back pain
The QUALEFFO-31 Questionnaire | up to 12 month
  The Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31), which contains three domains including pain, physical function, and mental function. This scale is assessed on a scale of 0 to 100, with 0 indicating the highest QoL and 100 the lowest
The EQ-5D Questionnaire | up to 12 month
  The EuroQol five-dimension (EQ-5D) questionnaire evaluates health status consisting five dimensions: mobility, selfcare, performance of usual activities, pain or discomfort, and anxiety or depression. After conversion, the index was between 0 and 1.0 (minimum score: 0, indicating worst health state; full score:1.0, indicating full health).
Secondary fracture rate | up to 12 month
  Secondary fracture rate containing vertebral fracture and non-vertebral fracture was assessed at 12 month after surgery. The lowest score was 0, the highest score was 100%. The lower score 0 represents no secondary fracture.
Adverse events | up to 12 month
  The main adverse events including deep venous thrombosis, pneumonia, acute renal failure, pulmonary embolism, myocardial infarction, influenza, transfer to intensive care unit, joint pain, headache, nausea, osteonecrosis of the jaw, atypical femoral fracture and rash.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No